CLINICAL TRIAL: NCT04699123
Title: The Study of NC318 Alone or in Combination With Pembrolizumab in Patients With Advanced Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NextCure, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Scott Gettinger, MD, Professor of Internal Medicine (Medical Oncology), Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000028206; 2P50CA196530-06 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2021-01-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1a - NC318 only (Experimental): At the discretion of the treating physician, advanced NSCLC patients on arm 1a will receive NC318 alone.
  Interventions: Drug: NC318 800 mg
- Arm 1b - NC318 and Pembrolizumab (Experimental): At the discretion of the treating physician, advanced NSCLC patients on arm 1b will receive combination therapy with NC318 and pembrolizumab.
  Interventions: Drug: NC318 400 mg; Drug: Pembrolizumab
- Arm 1c - NC318 and Pembrolizumab (Experimental): At the discretion of the treating physician, advanced NSCLC patients on arm 1b will receive combination therapy with NC318 and pembrolizumab.
  Interventions: Drug: NC318 800 mg
- Arm 2 (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab (Experimental): Arm 2 will enroll patients with advanced NSCLC who are naïve to PD-1 axis inhibitor therapy to receive therapy with NC318 in combination with pembrolizumab.
  Interventions: Drug: NC318 400 mg; Drug: Pembrolizumab
- Arm 2a (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab (Experimental): Arm 2a will enroll patients with advanced NSCLC who are naïve to PD-1 axis inhibitor therapy to receive combination therapy with NC318 and pembrolizumab.
  Interventions: Drug: NC318 800 mg; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NC318 800 mg — NC318 will be given intravenously (IV) weekly for 8 doses and then every 2 weeks for patients receiving combination therapy treatment or weekly for patient receiving NC318 in monotherapy.
  Arms: Arm 1a - NC318 only; Arm 1c - NC318 and Pembrolizumab; Arm 2a (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab
Drug: NC318 400 mg — NC318 will be given intravenously (IV) every 2 weeks.
  Arms: Arm 1b - NC318 and Pembrolizumab; Arm 2 (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab 200 mg will be given IV every 3 weeks
  Arms: Arm 1b - NC318 and Pembrolizumab; Arm 2 (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab; Arm 2a (naïve to PD-1 axis inhibitor)- NC318 and Pembrolizumab

SUMMARY:
This is a phase 2 study to investigate NC318 alone or in combination with Pembrolizumab in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a non-randomized, three-arm trial.

Arm 1a and 1b will enroll patients with advanced NSCLC regardless of tumor PD-L1 expression who have experienced disease progression on or after PD-1 axis inhibitor therapy, given alone or in combination with other systemic anti-cancer therapy. Patients will be assigned to arm 1a or 1b at the discretion of the treating physician. Patients on arm 1a will receive NC318 alone; those on arm 1b, combination therapy with NC318 and pembrolizumab.

Arm 1a will be based on a Simon two-stage minimax design. In the first stage, 18 patients will be accrued. If tumor response per RECIST v1.1 is achieved in 2 or fewer patients, arm 1a will be closed to further enrollment. If tumor response is demonstrated in 3 or more patients, then 25 additional patients will be accrued (stage 2), for a total of 43 patients.

Arm 1a and 1b will start with a safety run-in portion consisting of 6 patients (see 4.1.1). If deemed safe, each arm will continue to accrue and follow the Simon two-stage design outlined above. Patients in the run-in portion will be included in stage 1 of the Simon two-stage design.

Arm 2 will enroll patients with advanced NSCLC and tumor PD-L1 expression less than 50% who are naïve to PD-1 axis inhibitor therapy. Patients on arm 2 will receive combination therapy with NC318 and pembrolizumab. Arm 2 will also start with a safety run-in portion identical to that of arms 1a and 1b (see 4.1.1). If deemed safe, accrual will continue following a Simon two-stage minimax design. In the first stage, 19 patients will be accrued. If tumor response per RECIST v1.1 is achieved in 3 or fewer patients, arm 2 will be closed to further enrollment. If tumor response is demonstrated in 4 or more patients, then 36 additional patients will be accrued (stage 2), for a total of 54 patients. Patients in the run-in portion will be included in stage 1 of the Simon two-stage design.

The study protocol was amended to add 2 additional arms 5/2023. Arms 1c and 2a will receive NC318 800 mg, IV weekly for 8 doses, followed by every 2 week dosing. They both follow the same procedures as the earlier arms in the study. Arm 2 has essentially been removed from the study- but remains included in the protocol registration.

In addition, patients treated on arm 1a will be allowed to receive combination therapy with NC318 and pembrolizumab at the time of progression, after a mandatory tumor biopsy. They will be considered separately from arm 1c.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic (i.e., Stage IIIB not eligible for definitive chemoradiotherapy, Stage IV, or recurrent) NSCLC (per the American Joint Committee /AJCC staging system)
* ECOG performance status of 0 to 1
* Measurable disease per RECIST v1.1 criteria
* Arm 1a, and 1b and 1c: Prior PD-1 axis inhibitor therapy (anti-PD-1 or anti-PD-L1, e.g. nivolumab, pembrolizumab, atezolizumab, durvalumab, avelumab) either alone or in combination with other systemic agents, with documented progressive disease.
* Arm 2a: PD-L1 expression of less than 50 percent (PD-1 axis inhibitor therapy naïve)
* Patients with NSCLC known to harbor an ALK rearrangement, ROS1 rearrangement, EGFR mutation or BRAF mutation known to be sensitive to FDA approved tyrosine kinase inhibitors (TKI), are only eligible after experiencing disease progression (during or after treatment) or intolerance to respective TKI:

  1. Patients with TKI treated EGFR mutant NSCLC harboring the secondary EGFR T790M tumor must have received prior osimertinib.
  2. Patients with crizotinib treated ALK rearranged NSCLC must have received a next generation ALK inhibitor (e.g. ceritinib, alectinib, brigatinib or lorlatinib).
* At least one tumor amenable to incisional, excisional, core or forceps (transbronchial) biopsy. Patients must be willing to undergo a tumor biopsy before starting trial therapy and at the time of disease progression.
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Subjects must not have a history of life-threatening toxicity related to prior anti-PD-1 axis therapy:

  a. Subjects with history of anti-PD-1 axis therapy toxicities that are unlikely to recur with standard countermeasures (e.g., hormone replacement after adrenal crisis) are eligible.
* Symptomatic or untreated CNS metastases. Patients with a history of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  1. No evidence of interim progression between the completion of CNS-directed therapy and the start of trial therapy
  2. No ongoing requirement for dexamethasone as therapy for CNS disease; anticonvulsants at a stable dose are allowed.
  3. Completed stereotactic radiosurgery at least 1 week prior to initiation of trial therapyCycle 1, Day 1 or whole-brain radiation at least 2 weeks prior to initiation of trial therapyCycle 1, Day 1.
* History of leptomeningeal carcinomatosis
* Prior palliative radiotherapy outside the CNS within 2 weeks of the first dose of study drug
* Treatment with systemic immunosuppressive medications (including but not limited to, dexamethasone at doses > 2 mg daily (or equivalent dose of other corticosteroids), cyclophosphamide, tacrolimus, sirolimus, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor [anti-TNF] agents) within 2 weeks prior to initiating trial therapy. (Inhaled or topically applied steroids, and acute and chronic standard-dose NSAIDs are permitted. Replacement steroids are also permitted). Prophylactic corticosteroids prior to imaging with intravenous contrast are allowed per institutional guidelines, without need for delay of 2 weeks. Arm 2a: No prior PD-1 axis inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) in Arm 1a | Tumor response will be based on tumor assessments at screening, every 8 weeks from the first dose (for the first 24 weeks) and thereafter every 12 weeks until investigator-assessed initial disease progression, up to 4 years
  To determine the objective response rate (ORR) using RECIST v1.1 to NC318 in arm 1a
Objective response rate (ORR) in Arm 1b | Tumor response will be based on tumor assessments at screening, every 8 weeks from the first dose (for the first 24 weeks) and thereafter every 12 weeks until investigator-assessed initial disease progression, up to 4 years
  To determine the objective response rate (ORR) using RECIST v1.1 to NC318 combined with pembrolizumab in arm 1b
Objective response rate (ORR) in Arm 1c | Tumor response will be based on tumor assessments at screening, every 8 weeks from the first dose (for the first 24 weeks) and thereafter every 12 weeks until investigator-assessed initial disease progression, up to 4 years
  To determine the objective response rate (ORR) using RECIST v1.1 to NC318 combined with pembrolizumab in arm 1b
Number of participants on Arm 1b with treatment related adverse events as assessed by CTCAE v5 | Safety run in of 6 weeks
  To determine the safety of NC318 when administered in combination with pembrolizumab in arm 1b
Number of participants on Arm 1c with treatment related adverse events as assessed by CTCAE v5 | Safety run in of 6 weeks
  To determine the safety of NC318 when administered in combination with pembrolizumab in arm 1b
Objective response rate (ORR) in Arm 2 | Tumor response will be based on tumor assessments at screening, every 8 weeks from the first dose (for the first 24 weeks) and thereafter every 12 weeks until investigator-assessed initial disease progression, up to 4 years
  To determine the objective response rate (ORR) using RECIST v1.1 to NC318 combined with pembrolizumab in arm 2
Objective response rate (ORR) in Arm 2a | Tumor response will be based on tumor assessments at screening, every 8 weeks from the first dose (for the first 24 weeks) and thereafter every 12 weeks until investigator-assessed initial disease progression, up to 4 years
  To determine the objective response rate (ORR) using RECIST v1.1 to NC318 combined with pembrolizumab in arm 2
Number of participants in arm 2 with treatment related adverse events as assessed by CTCAE v5 | Safety run in of 6 weeks
  To determine the safety of NC318 when administered in combination with pembrolizumab in arm 2
Number of participants in arm 2a with treatment related adverse events as assessed by CTCAE v5 | Safety run in of 6 weeks
  To determine the safety of NC318 when administered in combination with pembrolizumab in arm 2

SECONDARY OUTCOMES:
Progression-free survival (RECIST v1.1) Arm 1a | Until disease progression or death, up to 4 years
  To determine progression-free survival (RECIST v1.1) with NC318 in patients with pre-treated advanced NSCLC who have experienced disease progression on or after anti-PD-1 axis therapy.
Overall Survival (RECIST v1.1) Arm 1a | Until death, up to 5 years
  To determine overall survival with NC318 in patients with pre-treated advanced NSCLC who have experienced disease progression on or after anti-PD-1 axis therapy.
Progression-free survival (RECIST v1.1) Arm 1B | Until disease progression or death, up to 4 years
  To determine progression-free survival (RECIST v1.1) with NC318 combined with pembrolizumab in patients with pre- treated advanced NSCLC who have experienced disease progression on or after anti-PD-1 axis therapy.
Overall survival (RECIST v1.1) Arm 1B | Until death, up to 5 years
  To determine overall survival (RECIST v1.1) with NC318 combined with pembrolizumab in patients with pre- treated advanced NSCLC who have experienced disease progression on or after anti-PD-1 axis therapy.
Progression-free survival (RECIST v1.1) Arm 2 | Until disease progression or death, up to 4 years
  To determine progression-free survival (RECIST v1.1) with NC318 and pembrolizumab when administered in combination to patients with PD-1 inhibitor naïve advanced NSCLC with tumor PD-L1 expression less than 50 percent.
Overall survival (RECIST v1.1) Arm 2 | Until death, up to 5 years
  To determine overall survival (RECIST v1.1) with NC318 and pembrolizumab when administered in combination to patients with PD-1 inhibitor naïve advanced NSCLC with tumor PD-L1 expression less than 50 percent.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gettinger, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No